CLINICAL TRIAL: NCT05426083
Title: Left Ventricular Physiological Effects of Veno-Arterial Extracorporeal Membrane Oxygenation Support During Cardiogenic Shock
Status: Recruiting | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: CV-2022-30951
Record Dates: First submitted 2022-06-15; First posted 2022-06-21 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Acute Coronary Syndrome; Cardiogenic Shock
Keywords: Acute Coronary Syndrome; Cardiogenic Shock; Left ventricle; VA-ECMO
MeSH Terms: conditions — Acute Coronary Syndrome; Shock, Cardiogenic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Physiological Assessment: Prospective physiological assessment of LV work and oxygen consumption in patients with SCAI D/E cardiogenic shock due to acute coronary syndrome treated with peripheral VA-ECMO support.
  Interventions: Other: Physiological Assessment

INTERVENTIONS:
Other: Physiological Assessment — Observational only

SUMMARY:
A Clinical Events Committee (CEC) will include Cardiac Surgery Professor and chief of cardiac surgery Rose Kelly MD, Professor of Medicine Ganesh Raveendran MD at the University of Minnesota who is the direction of Interventional Cardiology and Professor of Medicine at the University of Minnesota David Benditt. They will review and adjudicate serious and unexpected adverse events independently from the PI and co investigators.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years
* SCAI D/E CS requiring VA-ECMO support based on treating team's judgement.
* MAP >65 mmHg on <3 vasopressors/inotropes at the time of consent
* Cardiogenic shock due to acute coronary syndrome identified by coronary angiography at the index hospitalization per standard cardiology practice

Exclusion Criteria:

* VA-ECMO for sepsis, pulmonary embolism, COVID-19 related cardiorespiratory failure, severe RV failure due to severe idiopathic pulmonary hypertension
* CS due to other (non-ACS) etiologies
* Known patient with severe left ventricular dysfunction and stage IV NYHA heart failure being evaluated for or with a history of LVAD and transplantation prior to commencement of VA-ECMO
* Profound vasoplegia with MAP <65 mmHg on 3 vasopressors/inotropes
* Moderate to severe aortic regurgitation (contraindication to VA-ECMO)
* Moderate to severe aortic stenosis (contraindication to LV instrumentation with PV loop catheter)
* Bleeding complications requiring ongoing transfusions of blood products
* Ischemic lower extremities
* Evidence of circuit thrombosis or fibrin accumulation (turndown increases risk for stroke and clot formation)
* Evidence of sepsis or septic shock
* Evidence of LV thrombus on echocardiography (contraindication for accessing LV cavity with catheters)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients 18-75 years of age who were cannulated for VA-ECMO because of ischemic cardiogenic shock (SCAI shock categories D and E)44 per standard clinical practice. Acute coronary syndrome will be verified by the presence of an acute coronary cause identified on invasive coronary angiography.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-08-04 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Pressure-volume loops at the highest level of VA-ECMO support and the lowest level of VA-ECMO support. | Day 3 of ECMO
  Pressure-volume loops at the highest level of VA-ECMO support and the lowest level of VA-ECMO support.

CONTACTS AND LOCATIONS:
Overall Officials: Demetris Yannopoulous, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States